CLINICAL TRIAL: NCT02242643
Title: Immunogenicity and Safety Study of GSK Biologicals' Quadrivalent Influenza Vaccine (GSK2282512A) Compared to Fluzone® Quadrivalent in Children 6 to 35 Months of Age
Brief Title: Study to Evaluate the Immunogenicity and Safety of GlaxoSmithKline (GSK) Biologicals' Quadrivalent Influenza Vaccine (GSK2282512A) Compared to Fluzone® Quadrivalent in Children 6 to 35 Months of Age
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 201234
Record Dates: First submitted 2014-09-15; First posted 2014-09-17 (Estimated); Results first posted 2016-04-12 (Estimated); Last update posted 2018-09-07 (Actual); Status verified 2017-10

CONDITIONS: Influenza
Keywords: Fluzone Quadrivalent; Comparator; Children; Seasonal influenza; Safety; Immunogenicity
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor

ARMS (2):
- FluLaval™ Quadrivalent Group (Experimental): Subjects in this group received 1 dose (primed subjects) at Day 0 and 2 doses (unprimed subjects) at Days 0 and 28 of FluLaval™ Quadrivalent vaccine.
  The vaccine was administered intramuscularly into the anterolateral region of the thigh (subjects below 12 months of age) or in the deltoid muscle of the non-dominant arm (subjects ≥12 months of age).
  Interventions: Biological: FluLaval™ Quadrivalent
- Fluzone® Quadrivalent Group (Active Comparator): Subjects in this group received 1 dose (primed subjects) at Day 0 and 2 doses (unprimed subjects) at Days 0 and 28 of Fluzone® Quadrivalent vaccine.
  The vaccine was administered intramuscularly into the anterolateral region of the thigh (subjects below 12 months of age) or in the deltoid muscle of the non-dominant arm (subjects ≥12 months of age).
  Interventions: Biological: Fluzone® Quadrivalent

INTERVENTIONS:
Biological: FluLaval™ Quadrivalent — 1 or 2 doses administered intramusculary (IM) in deltoid region of non-dominant arm (for subjects ≥12 months of age) or anterolateral region of left thigh (for subjects <12 months of age) on Day 0 (primed subjects) and on Day 0 and Day 28 (unprimed subjects), respectively
  Other Names: FLU Q-QIV (GSK2282512A)
  Arms: FluLaval™ Quadrivalent Group
Biological: Fluzone® Quadrivalent — 1 or 2 doses administered IM in deltoid region of non-dominant arm (for subjects ≥12 months of age) or anterolateral region of left thigh (for subjects <12 months of age) on Day 0 (primed subjects) and on Day 0 and Day 28 (unprimed subjects), respectively
  Other Names: F-QIV
  Arms: Fluzone® Quadrivalent Group

SUMMARY:
The purpose of this study is to assess the immunogenicity and safety of GSK Biologicals' quadrivalent influenza vaccine (GSK2282512A) compared to Sanofi Pasteur's Fluzone® Quadrivalent in children 6 to 35 months of age.

ELIGIBILITY:
Inclusion Criteria:

* Subjects' parent(s)/Legally Acceptable Representative(s) [LAR(s)] who, in the opinion of the investigator, can and will comply with the requirements of the protocol.
* A male or female between, and including, 6 and 35 months of age at the time of the first vaccination.
* Written informed consent obtained from the parent(s)/LAR(s) of the subject.
* Subjects in stable health as determined by investigator's clinical examination and assessment of subject's medical history.
* Subjects are eligible regardless of history of administration of influenza vaccine in a previous season.

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine within 30 days preceding the first dose of study vaccine, or planned use during the study period. Routine registered childhood vaccinations are permitted.
* Child in care.
* Chronic administration (defined as more than 14 days in total) of immunosuppressants or other immune-modifying drugs within six months prior to the first vaccine dose. For corticosteroids, this will mean a dose equivalent to either > 2 mg/kg/day of body weight, or to ≥ 20 mg/day of prednisone for persons who weigh ≥ 10 kg, when administered for more than 2 weeks. Inhaled and topical steroids are allowed.
* Prior receipt of any seasonal or pandemic influenza vaccine (registered or investigational) within six months preceding the first dose of study vaccine, or planned use during the study period.
* Administration of immunoglobulins and/or any blood products within the three months preceding the first dose of study vaccine or planned administration during the study period.
* History of Guillain-Barré syndrome within six weeks of receipt of prior influenza vaccine.
* Any known or suspected allergy to any constituent of influenza vaccines (including egg proteins); a history of anaphylactic-type reaction to consumption of eggs; or a history of severe adverse reaction to a previous influenza vaccine.
* Acute disease and/or fever at the time of enrolment.

  * Fever is defined as temperature ≥ 38.0°C/100.4°F by any route.
  * Subjects with a minor illness (such as mild diarrhoea, mild upper respiratory infection) without fever may be enrolled at the discretion of the investigator.
* Any significant disorder of coagulation or treatment with warfarin derivatives or heparin.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* Any other condition which, in the opinion of the investigator, prevents the subject from participating in the study.

Ages: 6 Months to 35 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2432 (Actual)
Dates: Start 2014-10-01; Primary Completion 2015-03-16 (Actual); Study Completion 2015-06-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (61):
- United States (59):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Dothan, Alabama
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, Jonesboro, Arkansas
  - GSK Investigational Site, Anaheim, California
  - GSK Investigational Site, Chino, California
  - GSK Investigational Site, Daly City, California
  - GSK Investigational Site, Fresno, California
  - GSK Investigational Site, Hayward, California
  - GSK Investigational Site, Oakland, California
  - GSK Investigational Site, Paramount, California
  - GSK Investigational Site, Pleasanton, California
  - GSK Investigational Site, Sacramento, California
  - GSK Investigational Site, Santa Clara, California
  - GSK Investigational Site, Walnut Creek, California
  - GSK Investigational Site, West Covina, California
  - GSK Investigational Site, Colorado Springs, Colorado
  - GSK Investigational Site, Lake Mary, Florida
  - GSK Investigational Site, Miami Lakes, Florida
  - GSK Investigational Site, Nampa, Idaho
  - GSK Investigational Site, Augusta, Kansas
  - GSK Investigational Site, Newton, Kansas
  - GSK Investigational Site, Topeka, Kansas
  - GSK Investigational Site, Wichita, Kansas
  - GSK Investigational Site, Louisville, Kentucky
  - GSK Investigational Site, Bossier City, Louisiana
  - GSK Investigational Site, Metairie, Louisiana
  - GSK Investigational Site, Columbia, Maryland
  - GSK Investigational Site, Woburn, Massachusetts
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Lincoln, Nebraska
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Binghamton, New York
  - GSK Investigational Site, Syracuse, New York
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Beavercreek, Ohio
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Dayton, Ohio
  - GSK Investigational Site, Erie, Pennsylvania
  - GSK Investigational Site, Hermitage, Pennsylvania
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Sellersville, Pennsylvania
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Cheraw, South Carolina
  - GSK Investigational Site, Kingsport, Tennessee
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Fort Worth, Texas
  - GSK Investigational Site, Galveston, Texas
  - GSK Investigational Site, Tomball, Texas
  - GSK Investigational Site, Layton, Utah
  - GSK Investigational Site, Orem, Utah
  - GSK Investigational Site, Payson, Utah
  - GSK Investigational Site, Provo, Utah
  - GSK Investigational Site, Roy, Utah
  - GSK Investigational Site, Salt Lake City, Utah
  - GSK Investigational Site, South Jordan, Utah
  - GSK Investigational Site, Charlottesville, Virginia
  - GSK Investigational Site, Ellensburg, Washington
  - GSK Investigational Site, Marshfield, Wisconsin
- Mexico (2):
  - GSK Investigational Site, San Nicolás de los Garza, Nuevo León
  - GSK Investigational Site, Mexico City

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: 201234 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 201234 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 201234 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 201234 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 201234 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 201234 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 201234 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Primed subjects:Received atleast 2 doses of seasonal influenza vaccine since 1 July 2010 or atleast 1 dose of the 2013-2014 seasonal influenza vaccine. Unprimed subjects:Did not receive any seasonal influenza vaccine or received only 1 dose of seasonal influenza vaccine since 1 July 2010, but did not receive any 2013-2014 seasonal influenza vaccine
Pre-assignment Details: Data has been analyzed in sub-groups by age: 6-17 months and 18-35 months and by priming status.
  6 subjects were allocated subject numbers but did not receive the study vaccine dose and for 2 subjects the blood samples were withdrawn but they did not participate in the study due to screening failure.
Period: Overall Study
Arm/Group | FluLaval™ Quadrivalent Group | Fluzone® Quadrivalent Group
Started | 1207 | 1217
Completed | 1132 | 1139
Not Completed | 75 | 78
Not completed — Protocol Violation | 1 | 2
Not completed — Withdrawal by Subject | 15 | 10
Not completed — Migrated/moved from study area | 1 | 3
Not completed — Lost to Follow-up | 54 | 61
Not completed — Child placed in foster care by family | 0 | 1
Not completed — Non-compliance | 1 | 0
Not completed — Consent withdrawal by parent | 1 | 0
Not completed — Protocol requirements not followed | 1 | 0
Not completed — Language barrier | 1 | 0
Not completed — Withdrawal by subject at Visit 2 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FluLaval™ Quadrivalent Group | Fluzone® Quadrivalent Group | Total
Number analyzed (Participants) | 1207 | 1217 | 2424
Age, Continuous [Mean (Standard Deviation); unit: Months] | 19.4 (8.7) | 19.5 (8.9) | 19.45 (8.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 547 | 582 | 1129
  Male | 660 | 635 | 1295

OUTCOME MEASURES:

1. Primary Outcome: Haemagglutination Inhibition (HI) Antibody Titers Against Each of the 4 Vaccine Influenza Strains
Description: Antibody titers were expressed as Seroconversion rate (SCR) and SCR difference. SCR was defined as the proportion of vaccinees who had either a pre-vaccination titer < 1:10 and a post-vaccination titer ≥ 1:40 or a pre-vaccination titer ≥ 1:10 and at least a four-fold increase in post-vaccination titer.
  The vaccine strains assessed were Flu A/California/7/2009 (H1N1), A/Texas/50/2012 (H3N2), B/Massachusetts/2/2012 (Yamagata) and B/Brisbane/60/2008 (Victoria).
Time Frame: 28 days after last vaccine dose (i.e. Day 28 for vaccine-primed subjects and Day 56 for vaccine-unprimed subjects)
Population: The analysis was performed on the According-to-Protocol (ATP) cohort for immunogenicity which included all evaluable subjects, who received the study vaccine according to their treatment assignment and for whom the assay results for antibodies against at least one study vaccine strain after vaccination were available.
Measure: Number; unit: Subjects
Arm/Group | FluLaval™ Quadrivalent Group | Fluzone® Quadrivalent Group
Number analyzed (Participants) | 974 | 980
Subjects
  H1N1 [N=972,980] | 716 | 660
  H3N2 [N=972,980] | 740 | 680
  Victoria [N=973,980] | 631 | 475
  Yamagata [N=974,980] | 833 | 723
Statistical Analysis 1: Comparison: FluLaval™ Quadrivalent Group vs Fluzone® Quadrivalent Group; Test type: Non-Inferiority or Equivalence — Non-inferiority criterion: The upper limit of the two-sided 95% CI for the difference in SCR (Fluzone® Quadrivalent Group minus FluLaval™ Quadrivalent Group) did not exceed 10% for each of the four strains; Seroconversion rate (SCR) Difference (%) = -6.32, 95% CI 2-sided [-10.34 to -2.27] — For A/California/7/2009 (H1N1) vaccine strain
Statistical Analysis 2: Comparison: FluLaval™ Quadrivalent Group vs Fluzone® Quadrivalent Group; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; SCR Difference (%) = -6.74, 95% CI 2-sided [-10.68 to -2.80] — For A/Texas/50/2012 (H3N2) vaccine strain
Statistical Analysis 3: Comparison: FluLaval™ Quadrivalent Group vs Fluzone® Quadrivalent Group; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; SCR Difference (%) = -16.38, 95% CI 2-sided [-20.68 to -12.02] — For B/Massachusetts/2/2012 (Yamagata) vaccine strain
Statistical Analysis 4: Comparison: FluLaval™ Quadrivalent Group vs Fluzone® Quadrivalent Group; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; SCR Difference (%) = -11.75, 95% CI 2-sided [-15.28 to -8.21] — For B/Brisbane/60/2008 (Victoria) vaccine strain

2. Primary Outcome: Humoral Immune Response in Terms of Haemagglutination Inhibition (HI) Antibodies by Calculating Serum Antihaemagglutination (HA) Antibody Titers Against the 4 Vaccine Strains.
Description: HI antibody titres were expressed as geometric mean titers (GMTs) and adjusted GMT ratios. The vaccine strains assessed were Flu A/California/7/2009 (H1N1) HI, A/Texas/50/2012 (H3N2) HI, B/Massachusetts/2/2012 (Yamagata) HI and B/Brisbane/60/2008 (Victoria).
Time Frame: At 28 days after the last vaccine dose (i.e. Day 28 for vaccine-primed subjects and Day 56 for vaccine-unprimed subjects)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | FluLaval™ Quadrivalent Group | Fluzone® Quadrivalent Group
Number analyzed (Participants) | 1013 | 1028
Titers
  H1N1 | 98.8 [90.3 to 108.2] | 84.4 [76.9 to 92.6]
  H3N2 | 97.7 [90.3 to 105.7] | 84.3 [77.6 to 91.6]
  Yamagata | 257.5 [240.9 to 275.3] | 164.2 [151.8 to 177.6]
  Victoria | 55.1 [50.8 to 59.8] | 33.4 [30.6 to 36.4]
Statistical Analysis 1: Comparison: FluLaval™ Quadrivalent Group vs Fluzone® Quadrivalent Group; Test type: Non-Inferiority or Equivalence — Non-inferiority criterion: The upper limit of the two-sided 95% confidence interval (CI) for the GMT ratio (Fluzone® Quadrivalent Group/FluLaval™ Quadrivalent Group) did not exceed 1.5 for each of the four strains; Adjusted GMT ratio = 0.85, 95% CI 2-sided [0.77 to 0.95] — The GMTs were used to calculate the Adjusted GMTs, which in turn were used to calculate the Adjusted GMT ratio with 95% confidence interval (Ancova model: adjustment for baseline titer - pooled variance)
Statistical Analysis 2: Comparison: FluLaval™ Quadrivalent Group vs Fluzone® Quadrivalent Group; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Adjusted GMT Ratio = 0.85, 95% CI 2-sided [0.77 to 0.94] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: FluLaval™ Quadrivalent Group vs Fluzone® Quadrivalent Group; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Adjusted GMT Ratio = 0.65, 95% CI 2-sided [0.59 to 0.71] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 4: Comparison: FluLaval™ Quadrivalent Group vs Fluzone® Quadrivalent Group; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Adjusted GMT Ratio = 0.62, 95% CI 2-sided [0.56 to 0.69] — [estimate comment as in outcome 2, analysis 1]

3. Secondary Outcome: Haemagglutination Inhibition (HI) Antibody Titers Against Each of the 4 Vaccine Influenza Strains, Overall, by Age Group (6-17 and 18-35 Months of Age) and by Priming Status (Vaccine-primed and Vaccine-unprimed)
Description: Antibody titers were expressed as Geometric mean titers (GMTs). The vaccine strains assessed were A/California/7/2009 (H1N1), A/Texas/50/2012 (H3N2), B/Massachusetts/2/2012 (Yamagata) and B/Brisbane/60/2008 (Victoria).
Time Frame: At Day 0 and 28 days after last vaccine dose (i.e. Day 28 for vaccine-primed subjects and Day 56 for vaccine-unprimed subjects)
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Titers
Arm/Group | FluLaval™ Quadrivalent Group | Fluzone® Quadrivalent Group
Number analyzed (Participants) | 1013 | 1028
Titers
  H1N1, Day 0 | 11.0 [10.2 to 12.0] | 11.1 [10.2 to 12.0]
  H1N1, Day 28/Day 56 | 98.8 [90.3 to 108.2] | 84.4 [76.9 to 92.6]
  H3N2, Day 0 | 9.2 [8.6 to 9.8] | 9.6 [8.9 to 10.3]
  H3N2, Day 28/Day 56 | 97.7 [90.3 to 105.7] | 84.3 [77.6 to 91.6]
  Yamagata, Day 0 | 20.3 [18.8 to 22.0] | 20.6 [19.0 to 22.4]
  Yamagata, Day 28/Day 56 | 257.5 [240.9 to 275.3] | 164.2 [151.8 to 177.6]
  Victoria, Day 0 | 6.2 [6.0 to 6.5] | 6.3 [6.0 to 6.6]
  Victoria, Day 28/Day 56 | 55.1 [50.8 to 59.8] | 33.4 [30.6 to 36.4]
  H1N1, 6-17M, Day 0 | 7.2 [6.5 to 7.9] | 7.1 [6.5 to 7.7]
  H1N1, 6-17M, Day 28/Day 56 | 42.7 [37.1 to 49.0] | 43.2 [37.3 to 50.0]
  H1N1, 18-35M, Day 0 | 14.5 [13.0 to 16.2] | 14.6 [13.1 to 16.4]
  H1N1, 18-35M, Day 28/Day 56 | 170.9 [155.2 to 188.3] | 129.6 [116.3 to 144.3]
  H3N2, 6-17M, Day 0 | 5.8 [5.5 to 6.1] | 6.2 [5.8 to 6.7]
  H3N2, 6-17M, Day 28/Day 56 | 58.9 [52.2 to 66.4] | 54.8 [47.9 to 62.7]
  H3N2, 18-35M, Day 0 | 12.3 [11.1 to 13.6] | 12.5 [11.2 to 13.9]
  H3N2, 18-35M, Day 28/Day 56 | 136.0 [123.7 to 149.6] | 111.1 [100.6 to 122.7]
  Yamagata, 6-17M, Day 0 | 12.2 [11.1 to 13.5] | 13.0 [11.8 to 14.4]
  Yamagata, 6-17M, Day 28/Day 56 | 151.0 [137.4 to 165.9] | 79.1 [70.9 to 88.1]
  Yamagata, 18-35M, Day 0 | 28.0 [25.2 to 31.0] | 27.4 [24.5 to 30.7]
  Yamagata, 18-35M, Day 28/Day 56 | 364.8 [336.7 to 395.3] | 262.1 [239.3 to 287.1]
  Victoria, 6-17M, Day 0 | 5.5 [5.3 to 5.7] | 5.6 [5.3 to 5.9]
  Victoria, 6-17M, Day 28/Day 56 | 68.7 [61.8 to 76.3] | 31.9 [28.4 to 35.7]
  Victoria, 18-35M, Day 0 | 6.8 [6.4 to 7.3] | 6.8 [6.3 to 7.3]
  Victoria, 18-35M, Day 28/Day 56 | 47.8 [42.6 to 53.6] | 34.4 [30.4 to 38.8]
  H1N1, Unprimed, Day 0 | 7.5 [6.8 to 8.4] | 8.2 [7.4 to 9.2]
  H1N1, Unprimed, Day 56 | 51.4 [44.7 to 59.1] | 56.0 [48.4 to 64.8]
  H1N1, Primed, Day 0 | 14.4 [12.9 to 16.1] | 13.8 [12.3 to 15.4]
  H1N1, Primed, Day 28 | 158.8 [143.3 to 176.0] | 115.0 [102.6 to 128.9]
  H3N2, Unprimed, Day 0 | 6.4 [5.9 to 7.0] | 6.9 [6.3 to 7.6]
  H3N2, Unprimed, Day 56 | 75.0 [66.0 to 85.3] | 76.8 [66.9 to 88.3]
  H3N2, Primed, Day 0 | 11.8 [10.7 to 13.0] | 12.2 [10.9 to 13.5]
  H3N2, Primed, Day 28 | 118.4 [107.5 to 130.3] | 90.4 [81.8 to 100.0]
  Yamagata, Unprimed, Day 0 | 11.4 [10.3 to 12.6] | 12.4 [11.2 to 13.7]
  Yamagata, Unprimed, Day 56 | 179.8 [163.7 to 197.4] | 98.1 [88.1 to 109.3]
  Yamagata, Primed, Day 0 | 30.5 [27.6 to 33.8] | 30.1 [27.0 to 33.6]
  Yamagata, Primed, Day 28 | 334.3 [306.4 to 364.7] | 242.2 [219.1 to 267.7]
  Victoria, Unprimed, Day 0 | 5.6 [5.3 to 5.9] | 5.6 [5.3 to 6.0]
  Victoria, Unprimed, Day 56 | 91.7 [83.8 to 100.3] | 44.8 [40.1 to 50.0]
  Victoria, Primed, Day 0 | 6.7 [6.3 to 7.2] | 6.8 [6.4 to 7.3]
  Victoria, Primed, Day 28 | 38.1 [34.0 to 42.8] | 26.7 [23.6 to 30.3]

4. Secondary Outcome: Number of Subjects Who Were Seroprotected for Anti-HI Antibodies Against Each of the 4 Vaccine Influenza Strains, Overall, by Age Group (6-17 and 18-35 Months of Age) and by Priming Status (Vaccine-primed and Vaccine-unprimed)
Description: A seroprotected subject was defined as a vaccinated subject with a serum HI titer greater than or equal to (≥) 1:40. The vaccine strains assessed were Flu A/California/7/2009 (H1N1) HI, A/Texas/50/2012 (H3N2) HI, B/Massachusetts/2/2012 (Yamagata) HI and B/Brisbane/60/2008 (Victoria).
Time Frame: as for outcome 3
Population: The ATP cohort for immunogenicity included all evaluable subjects who received the study vaccine according to their treatment assignment and for whom the assay results for antibodies against at least one study vaccine strain after vaccination were available.
Measure: Number; unit: Subjects
Arm/Group | FluLaval™ Quadrivalent Group | Fluzone® Quadrivalent Group
Number analyzed (Participants) | 1013 | 1028
Subjects
  H1N1, Day 0 | 191 | 190
  H1N1, Day 28/56 | 814 | 775
  H3N2, Day 0 | 135 | 140
  H3N2, Day 28/56 | 833 | 800
  Yamagata, Day 0 | 324 | 336
  Yamagata, Day 28/56 | 983 | 911
  Victoria, Day 0 | 40 | 46
  Victoria, Day 28/56 | 669 | 512
  H1N1, 6-17M, Day 0 | 32 | 25
  H1N1, 6-17M, Day 28/Day 56 | 245 | 240
  H1N1, 18-35M, Day 0 | 159 | 165
  H1N1, 18-35M, Day 28/Day 56 | 569 | 535
  H3N2, 6-17M, Day 0 | 12 | 15
  H3N2, 6-17M, Day 28/Day 56 | 281 | 272
  H3N2, 18-35M, Day 0 | 123 | 125
  H3N2, 18-35M, Day 28/Day 56 | 552 | 528
  Yamagata, 6-17M, Day 0 | 64 | 70
  Yamagata, 6-17M, Day 28/Day 56 | 377 | 311
  Yamagata, 18-35M, Day 0 | 260 | 266
  Yamagata, 18-35M, Day 28/Day 56 | 606 | 600
  Victoria, 6-17M, Day 0 | 2 | 7
  Victoria, 6-17M, Day 28/Day 56 | 313 | 206
  Victoria, 18-35M, Day 0 | 38 | 39
  Victoria, 18-35M, Day 28/Day 56 | 356 | 306
  H1N1, Unprimed, Day 0 | 42 | 46
  H1N1, Unprimed, Day 56 | 282 | 294
  H1N1, Primed, Day 0 | 149 | 144
  H1N1, Primed, Day 28 | 532 | 481
  H3N2, Unprimed, Day 0 | 27 | 31
  H3N2, Unprimed, Day 56 | 321 | 330
  H3N2, Primed, Day 0 | 108 | 109
  H3N2, Primed, Day 28 | 512 | 470
  Yamagata, Unprimed, Day 0 | 65 | 80
  Yamagata, Unprimed, Day 56 | 407 | 362
  Yamagata, Primed, Day 0 | 259 | 256
  Yamagata, Primed, Day 28 | 576 | 549
  Victoria, Unprimed, Day 0 | 9 | 11
  Victoria, Unprimed, Day 56 | 379 | 277
  Victoria, Primed, Day 0 | 31 | 35
  Victoria, Primed, Day 28 | 290 | 235

5. Secondary Outcome: Number of Seroconverted Subjects for Anti-HA Antibodies Against Each of the 4 Vaccine Influenza Strains, Overall, by Age Group (6-17 and 18-35 Months of Age) and by Priming Status (Vaccine-primed and Vaccine-unprimed)
Description: A seroconverted subject was defined as a vaccinated subject with either a pre-vaccination titer less than (<) 1:10 and a post-vaccination titer ≥ 1:40, or a pre-vaccination titer ≥ 1:10 and at least a 4-fold increase in post-vaccination titer. The vaccine strains assessed were Flu A/California/7/2009 (H1N1) HI, A/Texas/50/2012 (H3N2) HI, B/Massachusetts/2/2012 (Yamagata) HI and B/Brisbane/60/2008 (Victoria).
Time Frame: 28 days after last vaccine dose (i.e. Day 28 for vaccine-primed subjects and Day 56 for vaccine-unprimed subjects)
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | FluLaval™ Quadrivalent Group | Fluzone® Quadrivalent Group
Number analyzed (Participants) | 974 | 980
Subjects
  H1N1 [N=972,980] | 716 | 660
  H3N2 [N=972,980] | 740 | 680
  Yamagata [N=974,980] | 833 | 723
  Victoria [N=973,980] | 631 | 475
  H1N1, 6-17M [N=376,375] | 220 | 216
  H1N1, 18-35M [N=596,605] | 496 | 444
  H3N2, 6-17M [N=376,375] | 260 | 250
  H3N2, 18-35M [N=596,605] | 480 | 430
  Yamagata, 6-17M [N=376,375] | 299 | 232
  Yamagata, 18-35M [N=598,605] | 534 | 491
  Victoria, 6-17M [N=376,375] | 291 | 189
  Victoria, 18-35M [N=597,605] | 340 | 286

6. Secondary Outcome: Mean Geometric Increase (MGI) for Haemagglutination Inhibition (HI) Antibody Titer Against Each of the 4 Vaccine Influenza Strains, Overall, by Age Group (6-17 and 18-35 Months of Age) and by Priming Status (Vaccine-primed and Vaccine-unprimed)
Description: MGI was defined as the fold increase in serum HI GMTs post-vaccination compared to pre-vaccination (Day 0). The vaccine strains assessed were Flu A/California/7/2009 (H1N1) HI, A/Texas/50/2012 (H3N2) HI, B/Massachusetts/2/2012 (Yamagata) HI and B/Brisbane/60/2008 (Victoria).
Time Frame: 28 days after last vaccine dose (i.e. Day 28 for vaccine-primed subjects and Day 56 for vaccine-unprimed subjects)
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: Fold increase
Arm/Group | FluLaval™ Quadrivalent Group | Fluzone® Quadrivalent Group
Number analyzed (Participants) | 974 | 980
Fold increase
  H1N1 [N=972,980] | 9.0 [8.4 to 9.7] | 7.7 [7.1 to 8.3]
  H3N2 [N=972,980] | 10.7 [10.0 to 11.6] | 8.9 [8.2 to 9.7]
  Yamagata [N=974,980] | 12.7 [11.7 to 13.7] | 8.1 [7.5 to 8.8]
  Victoria [N=973,980] | 8.7 [8.1 to 9.4] | 5.4 [5.0 to 5.8]
  H1N1, 6-17M [N=376,375] | 6.0 [5.3 to 6.8] | 6.1 [5.2 to 7.1]
  H1N1, 18-35M [N=596,605] | 11.7 [10.7 to 12.8] | 8.9 [8.1 to 9.8]
  H3N2, 6-17M [N=376,375] | 10.2 [9.0 to 11.6] | 8.8 [7.7 to 10.2]
  H3N2, 18-35M [N=596,605] | 11.1 [10.1 to 12.1] | 9.0 [8.2 to 9.9]
  Yamagata, 6-17M [N=376,375] | 12.3 [10.7 to 14.3] | 6.1 [5.3 to 7.0]
  Yamagata, 18-35M [N=598,605] | 12.9 [11.8 to 14.0] | 9.7 [8.9 to 10.6]
  Victoria, 6-17M [N=376,375] | 12.3 [11.0 to 13.8] | 5.7 [5.1 to 6.4]
  Victoria, 18-35M [N=597,605] | 7.0 [6.4 to 7.7] | 5.2 [4.7 to 5.7]
  H1N1, Unprimed [N=402,417] | 6.9 [6.1 to 7.8] | 6.8 [5.9 to 7.8]
  H1N1, Primed [N=570, 563] | 10.9 [10.0 to 12.0] | 8.5 [7.7 to 9.3]
  H3N2, Unprimed [N=402,417] | 11.8 [10.4 to 13.4] | 11.2 [9.7 to 12.9]
  H3N2, Primed [N=570, 563] | 10.0 [9.1 to 10.9] | 7.6 [6.9 to 8.3]
  Yamagata, Unprimed [N=402,417] | 16.0 [13.9 to 18.5] | 8.0 [6.9 to 9.3]
  Yamagata, Primed [N=572, 563] | 10.7 [9.9 to 11.6] | 8.2 [7.6 to 8.9]
  Victoria, Unprimed [N=402,417] | 16.2 [14.8 to 17.8] | 8.0 [7.2 to 8.8]
  Victoria, Primed [N=571, 563] | 5.6 [5.1 to 6.1] | 4.0 [3.6 to 4.4]

7. Secondary Outcome: Number of Subjects Reporting Any and Grade 3 Solicited Local Symptoms, Overall, by Age Group (6-17 and 18-35 Months of Age) and by Priming Status (Vaccine-primed and Vaccine-unprimed)
Description: Solicited local symptoms assessed were pain, redness and swelling. Any was defined as any solicited local symptom reported irrespective of intensity and all subjects reporting 'Yes' for solicited symptom occurred but with missing values for at least one day during the solicited period. Grade 3 pain = Cried when limb is moved/spontaneously painful. Grade 3 redness and swelling was greater than 100 millimeters (mm) i.e. >100mm.
Time Frame: During a 7-day (Day 0 - Day 6) follow-up period after each vaccination
Population: The analysis was performed on the Total Vaccinated cohort which included all subjects with at least one vaccine administration documented and for whom data were available.
Measure: Number; unit: Subjects
Arm/Group | FluLaval™ Quadrivalent Group | Fluzone® Quadrivalent Group
Number analyzed (Participants) | 1156 | 1151
Subjects
  Any Pain, Dose 1 [N=1151,1146] | 464 | 429
  Grade 3 Pain, Dose 1 [N=1151,1146] | 28 | 16
  Any Redness, Dose 1 [N=1151,1146] | 15 | 15
  Grade 3 Redness, Dose 1 [N=1151,1146] | 0 | 0
  Any Swelling, Dose 1 [N=1151,1146] | 11 | 5
  Grade 3 Swelling, Dose 1 [N=1151,1146] | 0 | 0
  Any Pain, Dose 2 [N=490,493] | 138 | 147
  Grade 3 Pain, Dose 2 [N=490,493] | 9 | 3
  Any Redness, Dose 2 [N=490,493] | 1 | 2
  Grade 3 Redness, Dose 2 [N=490,493] | 0 | 0
  Any Swelling, Dose 2 [N=490,493] | 0 | 0
  Grade 3 Swelling, Dose 2 [N=490,493] | 0 | 0
  Any Pain, Across doses [N=1156,1151] | 509 | 462
  Grade 3 Pain, Across doses [N=1156,1151] | 34 | 19
  Any Redness, Across doses [N=1156,1151] | 16 | 16
  Grade 3 Redness, Across doses [N=1156,1151] | 0 | 0
  Any Swelling, Across doses [N=1156,1151] | 11 | 5
  Grade 3 Swelling, Across doses [N=1156,1151] | 0 | 0
  Any Pain, 6-17M, Dose 1 [N=478,465] | 175 | 173
  Grade 3 Pain, 6-17M, Dose 1 [N=478,465] | 11 | 12
  Any Redness, 6-17M, Dose 1 [N=478,465] | 2 | 2
  Grade 3 Redness, 6-17M, Dose 1 [N=478,465] | 0 | 0
  Any Swelling, 6-17M, Dose 1 [N=478,465] | 4 | 0
  Grade 3 Swelling, 6-17M, Dose 1 [N=478,465] | 0 | 0
  Any Pain, 18-35M, Dose 1 [N=673,681] | 289 | 256
  Grade 3 Pain, 18-35M, Dose 1 [N=673,681] | 17 | 4
  Any Redness, 18-35M, Dose 1 [N=673,681] | 13 | 13
  Grade 3 Redness, 18-35M, Dose 1 [N=673,681] | 0 | 0
  Any Swelling, 18-35M, Dose 1 [N=673,681] | 7 | 5
  Grade 3 Swelling, 18-35M, Dose 1 [N=673,681] | 0 | 0
  Any Pain, 6-17M, Dose 2 [N=373,372] | 103 | 108
  Grade 3 Pain, 6-17M, Dose 2 [N=373,372] | 6 | 1
  Any Redness, 6-17M, Dose 2 [N=373,372] | 1 | 0
  Grade 3 Redness, 6-17M, Dose 2 [N=373,372] | 0 | 0
  Any Swelling, 6-17M, Dose 2 [N=373,372] | 0 | 0
  Grade 3 Swelling, 6-17M, Dose 2 [N=373,372] | 0 | 0
  Any Pain, 18-35M, Dose 2 [N=117,121] | 35 | 39
  Grade 3 Pain, 18-35M, Dose 2 [N=117,121] | 3 | 2
  Any Redness, 18-35M, Dose 2 [N=117,121] | 0 | 2
  Grade 3 Redness, 18-35M, Dose 2 [N=117,121] | 0 | 0
  Any Swelling, 18-35M, Dose 2 [N=117,121] | 0 | 0
  Grade 3 Swelling, 18-35M, Dose 2 [N=117,121] | 0 | 0
  Any Pain, 6-17M, Across Doses [N=481,469] | 211 | 196
  Grade 3 Pain, 6-17M, Across Doses [N=481,469] | 15 | 13
  Any Redness, 6-17M, Across Doses [N=481,469] | 3 | 2
  Grade 3 Redness, 6-17M, Across Doses [N=481,469] | 0 | 0
  Any Swelling, 6-17M, Across Doses [N=481,469] | 4 | 0
  Grade 3 Swelling, 6-17M, Across Doses [N=481,469] | 0 | 0
  Any Pain, 18-35M, Across Doses [N=675,682] | 298 | 266
  Grade 3 Pain, 18-35M, Across Doses [N=675,682] | 19 | 6
  Any Redness, 18-35M, Across Doses [N=675,682] | 13 | 14
  Grade 3 Redness, 18-35M, Across Doses [N=675,682] | 0 | 0
  Any Swelling, 18-35M, Across Doses [N=675,682] | 7 | 5
  Grade 3 Swelling, 18-35M, Across Doses [N=675,682] | 0 | 0
  Any Pain, Unprimed, Dose 1 [N=518,516] | 187 | 190
  Grade 3 Pain, Unprimed, Dose 1 [N=518,516] | 12 | 11
  Any Redness, Unprimed, Dose 1 [N=518,516] | 2 | 2
  Grade 3 Redness, Unprimed, Dose 1 [N=518,516] | 0 | 0
  Any Swelling, Unprimed, Dose 1 [N=518,516 | 4 | 0
  Grade 3 Swelling, Unprimed, Dose 1 [N=518,516] | 0 | 0
  Any Pain, Primed, Dose 1 [N=633,630] | 277 | 239
  Grade 3 Pain, Primed, Dose 1 [N=633,630] | 16 | 5
  Any Redness, Primed, Dose 1 [N=633,630] | 13 | 13
  Grade 3 Redness, Primed, Dose 1 [N=633,630] | 0 | 0
  Any Swelling, Primed, Dose 1 [N=633,630] | 7 | 5
  Grade 3 Swelling, Primed, Dose 1 [N=633,630] | 0 | 0
  Any Pain, Unprimed, Dose 2 [N=490,493] | 138 | 147
  Grade 3 Pain, Unprimed, Dose 2 [N=490,493] | 9 | 3
  Any Redness, Unprimed, Dose 2 [N=490,493] | 1 | 2
  Grade 3 Redness, Unprimed, Dose 2 [N=490,493] | 0 | 0
  Any Swelling, Unprimed, Dose 2 [N=490,493] | 0 | 0
  Grade 3 Swelling, Unprimed, Dose 2 [N=490,493] | 0 | 0
  Any Pain, Unprimed, Across Doses [N=523,521] | 232 | 223
  Grade 3 Pain, Unprimed, Across Doses [N=523,521] | 18 | 14
  Any Redness, Unprimed, Across Doses [N=523,521] | 3 | 3
  Grade 3 Redness, Unprimed, Across Doses[N=523,521] | 0 | 0
  Any Swelling, Unprimed, Across Doses [N=523,521] | 4 | 0
  Grade 3 Swelling,Unprimed, Across Doses[N=523,521] | 0 | 0
  Any Pain, Primed, Across Doses [N=633,630] | 277 | 239
  Grade 3 Pain, Primed, Across Doses [N=633,630] | 16 | 5
  Any Redness, Primed, Across Doses [N=633,630] | 13 | 13
  Grade 3 Redness, Primed, Across Doses [N=633,630] | 0 | 0
  Any Sweling, Primed, Across Doses [N=633,630] | 7 | 5
  Grade 3 Swelling, Primed, Across Doses [N=633,630] | 0 | 0

8. Secondary Outcome: Number of Subjects Reporting Any, Grade 3 and Related Solicited General Symptoms, Overall, by Age Group (6-17 and 18-35 Months of Age) and by Priming Status (Vaccine-primed and Vaccine-unprimed)
Description: Solicited general symptoms assessed were drowsiness, irritability/fussiness, loss of appetite and fever. Any was defined as any solicited general symptom reported irrespective of intensity and relationship to vaccination. Related was defined as symptoms assessed by the investigator to have a causal relationship to vaccination. Grade 3 irritability/fussiness was defined as crying that could not be comforted/prevented normal activity. Grade 3 loss of appetite was defined as not eating at all. Grade 3 drowsiness was defined as drowsiness that prevented normal activity. Any fever was defined as subjects with a documented temperature of greater than or equal to (≥) 38°C/100.4°F by any route and all subjects reporting temperature less than (< )38°C but with missing values for at least one day during the solicited period. Grade 3 fever was defined as temperature greater than (>) 39.0°C.
Time Frame: During the 7-day (Days 0-6) follow-up period after each vaccination
Population: as for outcome 7
Measure: Number; unit: Subjects
Arm/Group | FluLaval™ Quadrivalent Group | Fluzone® Quadrivalent Group
Number analyzed (Participants) | 1159 | 1152
Subjects
  Any Drowsiness, Dose 1 [N=1155,1148] | 424 | 424
  Grade 3 Drowsiness, Dose 1 [N=1155,1148] | 31 | 30
  Related Drowsiness, Dose 1 [N=1155,1148] | 365 | 381
  Any Fever, Dose 1 [N=1155,1148] | 146 | 147
  Fever (≥38.0°C), Dose 1 [N=1155,1148] | 65 | 67
  Grade 3 Fever, Dose 1 [N=1155,1148] | 16 | 11
  Related Fever, Dose 1 [N=1155,1148] | 41 | 50
  ≥38.0°C Related Fever, Dose 1 [N=1155,1148] | 41 | 50
  Any Irritability, Dose 1 [N=1155,1148] | 570 | 527
  Grade 3 Irritability, Dose 1 [N=1155,1148] | 44 | 34
  Related Irritability, Dose 1 [N=1155,1148] | 499 | 473
  Any Loss of Appetite, Dose 1 [N=1155,1148] | 334 | 328
  Grade 3 Loss of Appetite, Dose 1 [N=1155,1148] | 19 | 15
  Related Loss of Appetite, Dose 1 [N=1155,1148] | 280 | 290
  Any Drowsiness, Dose 2 [N=490,495] | 157 | 166
  Grade 3 Drowsiness, Dose 2 [N=490,495] | 10 | 6
  Related Drowsiness, Dose 2 [N=490,495] | 133 | 136
  Any Fever, Dose 2 [N=490,495] | 60 | 48
  Fever (≥38.0°C), Dose 2 [N=490,495] | 31 | 22
  Grade 3 Fever, Dose 2 [N=490,495] | 9 | 6
  Related Fever, Dose 2 [N=490,495] | 22 | 14
  ≥38.0°C Related Fever, Dose 2 [N=490,495] | 20 | 13
  Any Irritability, Dose 2 [N=490,495] | 211 | 214
  Grade 3 Irritability, Dose 2 [N=490,495] | 21 | 14
  Related Irritability, Dose 2 [N=490,495] | 185 | 175
  Any Loss of Appetite, Dose 2 [N=490,495] | 110 | 116
  Grade 3 Loss of Appetite, Dose 2 [N=490,495] | 8 | 5
  Related Loss of Appetite, Dose 2 [N=490,495] | 91 | 87
  Any Drowsiness, Across Doses [N=1159,1152] | 471 | 471
  Grade 3 Drowsiness, Across Doses [N=1159,1152] | 36 | 34
  Related Drowsiness, Across Doses [N=1159,1152] | 411 | 425
  Any Fever, Across Doses [N=1159,1152] | 183 | 178
  Fever (≥38.0°C), Across Doses [N=1159,1152 | 91 | 86
  Grade 3 Fever, Across Doses [N=1159,1152] | 25 | 17
  Related Fever, Across Doses [N=1159,1152] | 62 | 63
  ≥38.0°C Related Fever, Across Doses [N=1159,1152] | 60 | 62
  Any Irritability, Across Doses [N=1159,1152] | 630 | 582
  Grade 3 Irritability, Across Doses [N=1159,1152] | 61 | 45
  Related Irritability, Across Doses [N=1159,1152] | 558 | 525
  Any Loss of Appetite, Across Doses [N=1159,1152] | 391 | 385
  Grade 3 Loss of Appetite,Across Doses[N=1159,1152 | 26 | 19
  Related Loss of Appetite,Across Doses[N=1159,1152] | 328 | 337
  Any Drowsiness, 6-17M, Dose 1 [N=478,467] | 200 | 210
  Grade 3 Drowsiness, 6-17M, Dose 1 [N=478,467] | 16 | 17
  Related Drowsiness, 6-17M, Dose 1 [N=478,467] | 171 | 189
  Any Fever, 6-17M, Dose 1 [N=478,467] | 80 | 70
  Fever (≥38.0°C), 6-17M, Dose 1 [N=478,467] | 40 | 31
  Grade 3 Fever, 6-17M, Dose 1 [N=478,467] | 12 | 4
  Related Fever, 6-17M, Dose 1 [N=478,467] | 25 | 26
  ≥38.0°C Related Fever, 6-17M, Dose 1 [N=478,467] | 25 | 26
  Any Irritability, 6-17M, Dose 1 [N=478,467] | 273 | 252
  Grade 3 Irritability, 6-17M, Dose 1 [N=478,467] | 24 | 15
  Related Irritability, 6-17M, Dose 1 [N=478,467] | 239 | 227
  Any Loss of Appetite, 6-17M, Dose 1 [N=478,467] | 141 | 131
  Grade 3 Loss of Appetite, 6-17M,Dose 1 [N=478,467] | 7 | 4
  Related Loss of Appetite, 6-17M, Dose 1[N=478,467] | 122 | 115
  Any Drowsiness, 18-35M, Dose 1 [N=677,681] | 224 | 214
  Grade 3 Drowsiness, 18-35M, Dose 1 [N=677,681] | 15 | 13
  Related Drowsiness, 18-35M, Dose 1 [N=677,681] | 194 | 192
  Any Fever, 18-35M, Dose 1 [N=677,681] | 66 | 77
  Fever (≥38.0°C), 18-35M, Dose 1 [N=677,681] | 25 | 36
  Grade 3 Fever, 18-35M, Dose 1 [N=677,681] | 4 | 7
  Related Fever, 18-35M, Dose 1 [N=677,681] | 16 | 24
  ≥38.0°C Related Fever, 18-35M, Dose 1 [N=677,681] | 16 | 24
  Any Irritability, 18-35M, Dose 1 [N=677,681] | 297 | 275
  Grade 3 Irritability, 18-35M, Dose 1 [N=677,681] | 20 | 19
  Related Irritability, 18-35M, Dose 1 [N=677,681] | 260 | 246
  Any Loss of Appetite, 18-35M, Dose 1 [N=677,681] | 193 | 197
  Grade 3 Loss of Appetite,18-35M,Dose 1 [N=677,681] | 12 | 11
  Related Loss of Appetite,18-35M,Dose 1 [N=677,681] | 158 | 175
  Any Drowsiness, 6-17M, Dose 2 [N=373,374] | 129 | 142
  Grade 3 Drowsiness, 6-17M, Dose 2 [N=373,374] | 10 | 6
  Related Drowsiness, 6-17M, Dose 2 [N=373,374] | 111 | 115
  Any Fever, 6-17M, Dose 2 [N=373,374] | 47 | 38
  Fever (≥38.0°C), 6-17M, Dose 2 [N=373,374] | 23 | 16
  Grade 3 Fever, 6-17M, Dose 2 [N=373,374] | 5 | 3
  Related Fever, 6-17M, Dose 2 [N=373,374] | 17 | 11
  ≥38.0°C Related Fever, 6-17M, Dose 2 [N=373,374] | 15 | 10
  Any Irritability, 6-17M, Dose 2 [N=373,374] | 168 | 177
  Grade 3 Irritability, 6-17M, Dose 2 [N=373,374] | 16 | 12
  Related Irritability, 6-17M, Dose 2 [N=373,374] | 150 | 141
  Any Loss of Appetite, 6-17M, Dose 2 [N=373,374] | 90 | 91
  Grade 3 Loss of Appetite, 6-17M, Dose 2[N=373,374] | 8 | 3
  Related Loss of Appetite, 6-17M Dose 2[N=373,374] | 73 | 66
  Any Drowsiness, 18-35M, Dose 2 [N=117,121] | 28 | 24
  Grade 3 Drowsiness, 18-35M, Dose 2 [N=117,121] | 0 | 0
  Related Drowsiness, 18-35M, Dose 2 [N=117,121] | 22 | 21
  Any Fever, 18-35M, Dose 2 [N=117,121] | 13 | 10
  Fever (≥38.0°C), 18-35M, Dose 2 [N=117,121] | 8 | 6
  Grade 3 Fever, 18-35M, Dose 2 [N=117,121] | 4 | 3
  Related Fever, 18-35M, Dose 2 [N=117,121] | 5 | 3
  ≥38.0°C Related Fever, 18-35M, Dose 2 [N=117,121] | 5 | 3
  Any Irritability, 18-35M, Dose 2 [N=117,121] | 43 | 37
  Grade 3 Irritability, 18-35M, Dose 2 [N=117,121] | 5 | 2
  Related Irritability, 18-35M, Dose 2 [N=117,121] | 35 | 34
  Any Loss of Appetite, 18-35M, Dose 2 [N=117,121] | 20 | 25
  Grade 3 Loss of Appetite, 18-35M,Dose 2[N=117,121] | 0 | 2
  Related Loss of Appetite, 18-35M,Dose 2[N=117,121] | 18 | 21
  Any Drowsiness, 6-17M, Across Doses [N=481,470] | 238 | 248
  Grade 3 Drowsiness, 6-17M, Across Doses[N=481,470] | 21 | 21
  Related Drowsiness, 6-17M, Across Doses[N=481,470] | 209 | 224
  Any Fever, 6-17M, Across Doses [N=481,470] | 109 | 93
  Fever (≥38.0°C), 6-17M, Across Doses [N=481,470] | 60 | 45
  Grade 3 Fever, 6-17M, Across Doses [N=481,470] | 17 | 7
  Related Fever, 6-17M, Across Doses [N=481,470] | 41 | 36
  ≥38.0°CRelated Fever,6-17M,Across Doses[N=481,470] | 39 | 35
  Any Irritability, 6-17M, Across Doses [N=481,470] | 315 | 297
  Grade 3 Irritability,6-17M,Across Doses[N=481,470] | 36 | 25
  Related Irritability,6-17M,Across Doses[N=481,470] | 280 | 269
  Any Loss of Appetite,6-17M,Across Doses[N=481,470] | 188 | 175
  Grade3 LossofAppetite,6-17M,AcrossDoses[N=481,470] | 14 | 6
  Related LossofAppetite,6-17M,AcrossDoses[N=481,470 | 159 | 148
  Any Drowsiness, 18-35M, Across Doses [N=678,682] | 233 | 223
  Grade 3 Drowsiness,18-35M, Across Doses[N=678,682] | 15 | 13
  Related Drowsiness,18-35M,Across Doses [N=678,682] | 202 | 201
  Any Fever, 18-35M, Across Doses [N=678,682] | 74 | 85
  Fever (≥38.0°C), 18-35M, Across Doses [N=678,682] | 31 | 41
  Grade 3 Fever, 18-35M, Across Doses [N=678,682] | 8 | 10
  Related Fever, 18-35M, Across Doses [N=678,682] | 21 | 27
  ≥38.0°CRelated Fever,18-35M,Across Doses[N=678,682 | 21 | 27
  Any Irritability, 18-35M, Across Doses [N=678,682] | 315 | 285
  Grade3 Irritability,18-35M,Across Doses[N=678,682] | 25 | 20
  Related Irritability,18-35M,Across Doses[N=678,682 | 278 | 256
  Any Loss ofAppetite,18-35M,Across Doses[N=678,682] | 203 | 210
  Grade3LossofAppetite,18-35M,AcrossDoses[N=678,682] | 12 | 13
  RelatedLossofAppetite,18-35M,AcrossDoses[N=678,682 | 169 | 189
  Any Drowsiness, Unprimed, Dose 1 [N=520,518] | 212 | 211
  Grade 3 Drowsiness, Unprimed, Dose 1 [N=520,518] | 15 | 19
  Related Drowsiness, Unprimed, Dose 1 [N=520,518] | 182 | 189
  Any Fever, Unprimed, Dose 1 [N=520,518] | 80 | 69
  Fever (≥38.0°C), Unprimed, Dose 1 [N=520,518] | 41 | 33
  Grade 3 Fever, Unprimed, Dose 1 [N=520,518] | 12 | 3
  Related Fever, Unprimed, Dose 1 [N=520,518] | 24 | 25
  ≥38.0°C Related Fever, Unprimed, Dose 1[N=520,518] | 24 | 25
  Any Irritability, Unprimed, Dose 1 [N=520,518] | 274 | 256
  Grade 3 Irritability, Unprimed, Dose 1 [N=520,518] | 21 | 14
  Related Irritability, Unprimed, Dose 1 [N=520,518] | 240 | 227
  Any Loss of Appetite, Unprimed, Dose 1 [N=520,518] | 154 | 138
  Grade3 Loss of Appetite,Unprimed,Dose 1[N=520,518] | 7 | 6
  Related Loss of Appetite,Unprimed,Dose1[N=520,518] | 129 | 119
  Any Drowsiness, Primed, Dose 1 [N=635,630] | 212 | 213
  Grade 3 Drowsiness, Primed, Dose 1 [N=635,630] | 16 | 11
  Related Drowsiness, Primed, Dose 1 [N=635,630] | 183 | 192
  Any Fever, Primed, Dose 1 [N=635,630] | 66 | 78
  Fever (≥38.0°C) Primed, Dose 1 [N=635,630] | 24 | 34
  Grade 3 Fever, Primed, Dose 1 [N=635,630] | 4 | 8
  Related Fevers, Primed, Dose 1 [N=635,630] | 17 | 25
  ≥38.0°C Related Fever, Primed, Dose 1 [N=635,630] | 17 | 25
  Any Irritability, Primed, Dose 1 [N=635,630] | 296 | 271
  Grade 3 Irritability, Primed, Dose 1 [N=635,630] | 23 | 20
  Related Irritability, Primed, Dose 1 [N=635,630] | 259 | 246
  Any Loss of Appetite, Primed, Dose 1 [N=635,630] | 180 | 190
  Grade 3 Loss of Appetite, Primed,Dose 1[N=635,630] | 12 | 9
  Related Loss of Appetite,Primed,Dose 1 [N=635,630] | 151 | 171
  Any Drowsiness, Unprimed, Dose 2 [N=490,495] | 157 | 166
  Grade 3 Drowsiness, Unprimed, Dose 2 [N=490,495] | 10 | 6
  Related Drowsiness, Unprimed, Dose 2 [N=490,495] | 133 | 136
  Any Fever, Unprimed, Dose 2 [N=490,495] | 60 | 48
  Fever (≥38.0°C), Unprimed, Dose 2 [N=490,495] | 31 | 22
  Grade 3 Fever, Unprimed, Dose 2 [N=490,495] | 9 | 6
  Related Fever, Unprimed, Dose 2 [N=490,495] | 22 | 14
  ≥38.0°C Related Fever, Unprimed,Dose 2 [N=490,495] | 20 | 13
  Any Irritability, Unprimed, Dose 2 [N=490,495] | 211 | 214
  Grade 3 Irritability, Unprimed, Dose 2 [N=490,495] | 21 | 14
  Related Irritability, Unprimed,Dose 2 [N=490,495] | 185 | 175
  Any Loss of Appetite, Unprimed, Dose 2 [N=490,495] | 110 | 116
  Grade3 Loss of Appetite,Unprimed,Dose 2[N=490,495] | 8 | 5
  Related Loss of Appetite,Unprimed,Dose 2[N=490,495 | 91 | 87
  Any Drowsiness, Unprimed, Across Doses [N=524,522] | 259 | 258
  Grade3 Drowsiness,Unprimed,Across Doses[N=524,522] | 20 | 23
  RelatedDrowsiness,Unprimed,Across Doses[N=524,522] | 228 | 233
  Any Fever, Unprimed, Across Doses [N=524,522] | 117 | 100
  Fever (≥38.0°C), Unprimed,Across Doses [N=524,522] | 67 | 52
  Grade 3 Fever, Unprimed, Across Doses [N=524,522] | 21 | 9
  Related Fever, Unprimed, Across Doses [N=524,522] | 45 | 38
  ≥38.0°CRelatedFever,Unprimed,AcrossDoses[N=524,522 | 43 | 37
  Any Irritability,Unprimed, Across Doses[N=524,522] | 334 | 311
  Grade3Irritability,Unprimed,AcrossDoses[N=524,522] | 38 | 25
  RelatedIrritability,Unprimed,AcrossDoses[N=524,522 | 299 | 279
  AnyLoss ofAppetite,Unprimed,AcrossDoses[N=524,522] | 211 | 195
  Grade3LossofAppetite,Unprimed,AcrossDosesN=524,522 | 14 | 10
  RelatedLossofAppetite,UnprimedAcrossDosesN=524,522 | 177 | 166
  Any Drowsiness, Primed, Across Doses [N=635,630] | 212 | 213
  Grade 3 Drowsiness, Primed,Across Doses[N=635,630] | 16 | 11
  Related Drowsiness,Primed,Across Doses[N=635,630] | 183 | 192
  Any Fever, Primed, Across Doses [N=635,630] | 66 | 78
  Fever (≥38.0°C), Primed, Across Doses [N=635,630] | 24 | 34
  Grade 3 Fever, Primed, Across Doses [N=635,630] | 4 | 8
  Related Fever, Primed, Across Doses [N=635,630] | 17 | 25
  ≥38.0°C RelatedFever,Primed,Across Doses[N=635,630 | 17 | 25
  Any Irritability, Primed, Across Doses [N=635,630] | 296 | 271
  Grade3 Irritability,Primed,Across Doses[N=635,630] | 23 | 20
  Related Irritability,Primed,AcrossDoses[N=635,630] | 259 | 246
  Any Loss of Appetite,Primed,AcrossDoses[N=635,630] | 180 | 190
  Grade3 LossofAppetite,Primed,AcrossDoses[N=635,630 | 12 | 9
  RelatedLossofAppetite,Primed,AcrossDoses[N=635,630 | 151 | 171

9. Secondary Outcome: Duration of Solicited Local and General AEs, Overall, by Age Group (6-17 and 18-35 Months of Age) and by Priming Status (Vaccine-primed and Vaccine-unprimed)
Description: Duration was defined as number of days with any grade of local and general symptoms.
Time Frame: During the 7-day (Days 0-6) follow-up period after each vaccination.
Population: as for outcome 7
Measure: Median (Full Range); unit: Days
Arm/Group | FluLaval™ Quadrivalent Group | Fluzone® Quadrivalent Group
Number analyzed (Participants) | 570 | 527
Days
  Drowsiness, Dose 1 [N=424,424] | 1.0 [1.0 to 7.0] | 1.5 [1.0 to 7.0]
  Drowsiness, Dose 2 [N=157,166] | 2.0 [1.0 to 7.0] | 2.0 [1.0 to 7.0]
  Irritability, Dose 1 [N=570, 527] | 2.0 [1.0 to 7.0] | 2.0 [1.0 to 7.0]
  Irritability, Dose 2 [N=211,214] | 2.0 [1.0 to 7.0] | 2.0 [1.0 to 7.0]
  Loss of Appetite, Dose 1 [N=334, 328] | 2.0 [1.0 to 7.0] | 2.0 [1.0 to 7.0]
  Loss of Appetite, Dose 2 [N=110,116] | 2.0 [1.0 to 7.0] | 2.0 [1.0 to 7.0]
  Pain, Dose 1 [N=464,429] | 1.0 [1.0 to 7.0] | 2.0 [1.0 to 6.0]
  Pain, Dose 2 [N=138,147] | 1.0 [1.0 to 6.0] | 1.0 [1.0 to 5.0]
  Redness, Dose 1 [N=15,15] | 2.0 [1.0 to 4.0] | 1.0 [1.0 to 6.0]
  Redness, Dose 2 [N=1,2] | 1.0 [1.0 to 1.0] | 1.5 [1.0 to 2.0]
  Swelling, Dose 1 [N=11,5] | 2.0 [1.0 to 5.0] | 2.0 [1.0 to 3.0]
  Fever, Dose 1 [N=146,147] | 1.0 [1.0 to 7.0] | 1.0 [1.0 to 7.0]
  Fever, Dose 2 [N=60,48] | 1.0 [1.0 to 7.0] | 2.0 [1.0 to 7.0]
  Drowsiness, 6-17M, Dose 1 [N=200,210] | 2.0 [1.0 to 7.0] | 2.0 [1.0 to 7.0]
  Drowsiness, 18-35M, Dose 1 [N=224,214] | 1.0 [1.0 to 7.0] | 1.0 [1.0 to 7.0]
  Drowsiness, 6-17M, Dose 2 [N=129,142] | 2.0 [1.0 to 7.0] | 2.0 [1.0 to 7.0]
  Drowsiness, 18-35M, Dose 2 [N=28,24] | 2.0 [1.0 to 7.0] | 1.0 [1.0 to 4.0]
  Irritability, 6-17M, Dose 1 [N=273,252] | 2.0 [1.0 to 7.0] | 2.0 [1.0 to 7.0]
  Irritability, 18-35M, Dose 1 [N=297,275] | 2.0 [1.0 to 7.0] | 2.0 [1.0 to 7.0]
  Irritability, 6-17M, Dose 2 [N=168,177] | 2.0 [1.0 to 7.0] | 2.0 [1.0 to 7.0]
  Irritability, 18-35M, Dose 2 [N=43,37] | 2.0 [1.0 to 7.0] | 1.0 [1.0 to 7.0]
  Loss of Appetite, 6-17M, Dose 1 [N=141,131] | 2.0 [1.0 to 7.0] | 2.0 [1.0 to 7.0]
  Loss of Appetite, 18-35M, Dose 1 [N=193,197] | 2.0 [1.0 to 7.0] | 2.0 [1.0 to 7.0]
  Loss of Appetite, 6-17M, Dose 2 [N=90,91] | 2.0 [1.0 to 7.0] | 2.0 [1.0 to 7.0]
  Loss of Appetite, 18-35M, Dose 2 [N=20,25] | 2.0 [1.0 to 7.0] | 2.0 [1.0 to 7.0]
  Pain, 6-17M, Dose 1 [N=175,173] | 1.0 [1.0 to 7.0] | 1.0 [1.0 to 6.0]
  Pain, 18-35M, Dose 1 [N=289,256] | 2.0 [1.0 to 7.0] | 2.0 [1.0 to 6.0]
  Pain, 6-17M, Dose 2 [N=103,108] | 1.0 [1.0 to 6.0] | 2.0 [1.0 to 5.0]
  Pain, 18-35M, Dose 2 [N=35,39] | 1.0 [1.0 to 5.0] | 1.0 [1.0 to 4.0]
  Redness, 6-17M, Dose 1 [N=2,2] | 1.5 [1.0 to 2.0] | 1.0 [1.0 to 1.0]
  Redness, 18-35M, Dose 1 [N=13,13] | 2.0 [1.0 to 4.0] | 1.0 [1.0 to 6.0]
  Redness, 6-17M, Dose 2 [N=1,0] | 1.0 [1.0 to 1.0] | 0.0 [0.0 to 0.0]
  Redness, 18-35M, Dose 2 [N=0,2] | 0.0 [0.0 to 0.0] | 1.5 [1.0 to 2.0]
  Swelling, 6-17M, Dose 1 [N=4,0] | 1.5 [1.0 to 2.0] | 0.0 [0.0 to 0.0]
  Swelling, 18-35M, Dose 1 [N=7,5] | 2.0 [1.0 to 5.0] | 2.0 [1.0 to 3.0]
  Fever, 6-17M, Dose 1 [N=80,70] | 2.0 [1.0 to 7.0] | 1.0 [1.0 to 7.0]
  Fever, 18-35M, Dose 1 [N=66,77] | 1.0 [1.0 to 6.0] | 1.0 [1.0 to 6.0]
  Fever, 6-17M, Dose 2 [N=47,38] | 1.0 [1.0 to 7.0] | 1.5 [1.0 to 7.0]
  Fever, 18-35M, Dose 2 [N=13,10] | 1.0 [1.0 to 3.0] | 2.0 [1.0 to 3.0]
  Drowsiness, Unprimed, Dose 1 [N=212,211] | 2.0 [1.0 to 7.0] | 2.0 [1.0 to 7.0]
  Drowsiness, Primed, Dose 1 [N=212,213] | 1.0 [1.0 to 7.0] | 1.0 [1.0 to 7.0]
  Drowsiness, Unprimed, Dose 2 [N=157,166] | 2.0 [1.0 to 7.0] | 2.0 [1.0 to 7.0]
  Irritability, Unprimed, Dose 1 [N=274,256] | 2.0 [1.0 to 7.0] | 2.0 [1.0 to 7.0]
  Irritability, Primed, Dose 1 [N=296,271] | 2.0 [1.0 to 7.0] | 2.0 [1.0 to 7.0]
  Irritability, Unprimed, Dose 2 [N=211,214] | 2.0 [1.0 to 7.0] | 2.0 [1.0 to 7.0]
  Loss of Appetite, Unprimed, Dose 1 [N=154,138] | 2.0 [1.0 to 7.0] | 2.0 [1.0 to 7.0]
  Loss of Appetite, Primed, Dose 1 [N=180,190] | 1.0 [1.0 to 7.0] | 2.0 [1.0 to 7.0]
  Loss of Appetite, Unprimed, Dose 2 [N=110,116] | 2.0 [1.0 to 7.0] | 2.0 [1.0 to 7.0]
  Pain, Unprimed, Dose 1 [N=187,190] | 1.0 [1.0 to 7.0] | 1.0 [1.0 to 6.0]
  Pain, Primed, Dose 1 [N=277,239] | 2.0 [1.0 to 7.0] | 2.0 [1.0 to 6.0]
  Pain, Unprimed, Dose 2 [N=138,147] | 1.0 [1.0 to 6.0] | 1.0 [1.0 to 5.0]
  Redness, Unprimed, Dose 1 [N=2,2] | 1.5 [1.0 to 2.0] | 2.0 [1.0 to 3.0]
  Redness, Primed, Dose 1 [N=13,13] | 2.0 [1.0 to 4.0] | 1.0 [1.0 to 6.0]
  Redness, Unprimed, Dose 2 [N=1,2] | 1.0 [1.0 to 1.0] | 1.5 [1.0 to 2.0]
  Swelling, Unprimed, Dose 1 [N=4,0] | 1.5 [1.0 to 2.0] | 0.0 [0.0 to 0.0]
  Swelling, Primed, Dose 1 [N=7,5] | 2.0 [1.0 to 5.0] | 2.0 [1.0 to 3.0]
  Fever, Unprimed, Dose 1 [N=80,69] | 1.0 [1.0 to 7.0] | 1.0 [1.0 to 7.0]
  Fever, Primed, Dose 1 [N=66,78] | 1.0 [1.0 to 7.0] | 1.0 [1.0 to 6.0]
  Fever, Unprimed, Dose 2 [N=60,48] | 1.0 [1.0 to 7.0] | 2.0 [1.0 to 7.0]

10. Secondary Outcome: Number of Subjects Reporting Any Fever Following Each Dose and Across Doses.
Description: Any Fever = all subjects with a documented temperature of ≥38.0°C /100.4°F by axillary route and all subjects reporting temperature < 38.0°C but with missing values for at least one day during the solicited period.
  Grade 3 fever was defined as temperature greater than (>) 39.0°C.
Time Frame: During a 2-day (Days 0-1) follow-up period after each vaccination
Population: as for outcome 7
Measure: Number; unit: Subjects
Arm/Group | FluLaval™ Quadrivalent Group | Fluzone® Quadrivalent Group
Number analyzed (Participants) | 1159 | 1152
Subjects
  Any Fever, Dose 1 [N=1155,1148] | 63 | 74
  Fever (≥38.0°C), Dose 1 [N=1155,1148] | 30 | 34
  Grade 3 Fever (>39.0°C), Dose 1 [N=1155,1148] | 6 | 4
  Any Fever, Dose 2 [N=490,495] | 21 | 22
  Fever (≥38.0°C), Dose 2 [N=490,495] | 12 | 10
  Grade 3 Fever (>39.0°C), Dose 2 [N=490,495] | 3 | 2
  Any Fever, Across Doses [N=1159,1152] | 82 | 93
  Fever (≥38.0°C), Across Doses [N=1159,1152] | 42 | 43
  Grade 3 Fever (>39.0°C), Across Doses[N=1159,1152] | 9 | 6

11. Secondary Outcome: Number of Subjects Reporting the Occurrence of All Medically Attended Events (MAEs), Overall, by Age Group (6-17 and 18-35 Months of Age) and by Priming Status (Vaccine-primed and Vaccine-unprimed).
Description: MAEs were defined as adverse events with medically-attended visits that were not routine visits for physical examination or vaccination, such as visits for hospitalization, an emergency room visit, or an otherwise unscheduled visit to or from medical personnel (medical doctor) for any reason. Any was defined as any occurrence of MAE(s).
Time Frame: During the entire study period (Days 0 -180)
Population: as for outcome 7
Measure: Number; unit: Subjects
Arm/Group | FluLaval™ Quadrivalent Group | Fluzone® Quadrivalent Group
Number analyzed (Participants) | 1207 | 1217
Subjects
  Any MAE(s) [N=1207,1217] | 727 | 719
  Any MAE(s), 6-17M [N=500,502] | 322 | 323
  Any MAE(s), 18-35M [N=707,715] | 405 | 396
  Any MAE(s), Unprimed [N=550,560] | 344 | 337
  Any MAE(s), Primed [N=657,657] | 383 | 382

12. Secondary Outcome: Number of Subjects Reporting the Occurrence of Any and Related Potential Immune-Mediated Disease (pIMDs), Overall, by Age Group (6-17 and 18-35 Months of Age) and by Priming Status (Vaccine-primed and Vaccine-unprimed)
Description: pIMDs are a subset of adverse events (AEs) that include both clearly autoimmune diseases and also other inflammatory and/or neurologic disorders which may or may not have an autoimmune etiology. Related = symptom assed by the investigator as causally related to the study vaccination.
Time Frame: During the entire study period (Days 0 -180)
Population: as for outcome 7
Measure: Number; unit: Subjects
Arm/Group | FluLaval™ Quadrivalent Group | Fluzone® Quadrivalent Group
Number analyzed (Participants) | 1207 | 1217
Subjects
  Any pIMD(s) [N=1207,1217] | 1 | 1
  Related pIMD(s) [N=1207,1217] | 0 | 0
  Any pIMD(s), 6-17M [N=500,502] | 1 | 1
  Related pIMD(s), 6-17M [N=500,502] | 0 | 0
  Any pIMD(s), 18-35M [N=707,715] | 0 | 0
  Related pIMD(s), 18-35M [N=707,715] | 0 | 0
  Any pIMD(s), Unprimed [N=550,560] | 0 | 0
  Related pIMD(s), Unprimed [N=550,560] | 0 | 0
  Any pIMD(s), Primed [N=657,657] | 1 | 1
  Related pIMD(s), Primed [N=657,657] | 0 | 0

13. Secondary Outcome: Number of Subjects Reporting Any, Grade 3 and Related Unsolicited Adverse Events (AEs), Overall, by Age Group (6-17 and 18-35 Months of Age) and by Priming Status (Vaccine-primed and Vaccine-unprimed)
Description: An unsolicited AE was defined as an untoward medical occurrence in a patient or clinical investigation subject, temporally associated with use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as occurrence of any unsolicited symptom regardless of intensity grade or relation to vaccination. Grade 3 unsolicited AE was defined as an event that prevented normal activity. Related unsolicited AE was defined as an event assessed by the investigator to be causally related to the study vaccination.
Time Frame: During a 28-day (Days 0-27 for primed and unprimed subjects and Days 28-56 for unprimed subjects) post-vaccination period
Population: as for outcome 7
Measure: Number; unit: Subjects
Arm/Group | FluLaval™ Quadrivalent Group | Fluzone® Quadrivalent Group
Number analyzed (Participants) | 1207 | 1217
Subjects
  Any Unsolicited AEs [N=1207,1217] | 549 | 537
  Grade 3 Unsolicited AEs [N=1207,1217] | 70 | 75
  Related Unsolicited AEs [N=1207,1217] | 71 | 71
  Any Unsolicited AEs, 6-17M [N=500,502] | 268 | 270
  Grade 3 Unsolicited AEs, 6-17M [N=500,502] | 32 | 48
  Related Unsolicited AEs, 6-17M [N=500,502] | 36 | 33
  Any Unsolicited AEs, 18-35M [N=707,715] | 281 | 267
  Grade 3 Unsolicited AEs, 18-35M [N=707,715] | 38 | 27
  Related Unsolicited AEs, 18-35M [N=707,715] | 35 | 38
  Any Unsolicited AEs, Unprimed [N=550,560] | 310 | 302
  Grade 3 Unsolicited AEs, Unprimed [N=550,560] | 35 | 48
  Related Unsolicited AEs, Unprimed [N=550,560] | 40 | 35
  Any Unsolicited AEs, Primed [N=657,657] | 239 | 235
  Grade 3 Unsolicited AEs, Primed [N=657,657] | 35 | 27
  Related Unsolicited AEs, Primed [N=657,657] | 31 | 36

14. Secondary Outcome: Number of Subjects Reporting Any and Related Serious Adverse Events (SAEs), Overall, by Age Group (6-17 and 18-35 Months of Age) and by Priming Status (Vaccine-primed and Vaccine-unprimed)
Description: SAEs assessed include medical occurrences that results in death, are life threatening, require hospitalization or prolongation of hospitalization, results in disability/incapacity or are a congenital anomaly/birth defect in the offspring of a study subjects. Related = symptom assessed by the investigator as causally related to the study vaccination.
Time Frame: During the entire study period (Days 0 -180)
Population: as for outcome 7
Measure: Number; unit: Subjects
Arm/Group | FluLaval™ Quadrivalent Group | Fluzone® Quadrivalent Group
Number analyzed (Participants) | 1207 | 1217
Subjects
  Any SAE(s) [N=1207,1217] | 22 | 21
  Related SAE(s) [N=1207,1217] | 0 | 0
  Any SAE(s), 6-17M [N=500,502] | 11 | 11
  Related SAE(s), 6-17M [N=500,502] | 0 | 0
  Any SAE(s), 18-35M [N=707,715] | 11 | 10
  Related SAE(s), 18-35M [N=707,715] | 0 | 0
  Any SAE(s), Unprimed [N=550,560] | 8 | 13
  Related SAE(s), Unprimed [N=550,560] | 0 | 0
  Any SAE(s), Primed [N=657,657] | 14 | 8
  Related SAE(s), Primed [N=657,657] | 0 | 0

ADVERSE EVENTS:
Time Frame: Serious Adverse Events: From Day 0 to Day 180; Solicited local and general symptoms: During the 7-day (Days 0-6) post-vaccination period across doses; Unsolicited adverse events: During the 28-day post-vaccination period.
Description: For the systematically assessed other (non-serious) adverse events, the number of participants at risk included those from Total Vaccinated Cohort who had the symptom sheet completed.
Arm/Group | FluLaval™ Quadrivalent Group | Fluzone® Quadrivalent Group
Serious Adverse Events (participants affected / at risk) | 5/1207 | 4/1217
Other Adverse Events (participants affected / at risk) | 932/1207 | 895/1217
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | FluLaval™ Quadrivalent Group (N=1207) | Fluzone® Quadrivalent Group (N=1217)
Febrile convulsion (Nervous system disorders) | 5 | 4
Dehydration (Metabolism and nutrition disorders) | 2 | 3
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Bronchiolitis (Infections and infestations) | 1 | 2
Gastroenteritis (Infections and infestations) | 1 | 2
Cellulitis (Infections and infestations) | 1 | 1
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 2 | 0
Urinary tract infection (Infections and infestations) | 1 | 1
Abscess (Infections and infestations) | 0 | 1
Accidental exposure to product (Injury, poisoning and procedural complications) | 1 | 0
B precursor type acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Calculus urinary (Renal and urinary disorders) | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 | 0
Croup infectious (Infections and infestations) | 1 | 0
Developmental delay (General disorders) | 0 | 1
Failure to thrive (Metabolism and nutrition disorders) | 0 | 1
Gastroenteritis rotavirus (Infections and infestations) | 0 | 1
Groin abscess (Infections and infestations) | 1 | 0
Hemiplegia (Nervous system disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Intussusception (Gastrointestinal disorders) | 0 | 1
Kawasaki's disease (Vascular disorders) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Multiple injuries (Injury, poisoning and procedural complications) | 1 | 0
Otitis media acute (Infections and infestations) | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory syncytial virus infection (Infections and infestations) | 0 | 1
Seizure (Nervous system disorders) | 0 | 1
Sexual abuse (Social circumstances) | 1 | 0
Staphylococcal abscess (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | FluLaval™ Quadrivalent Group (N=1207) | Fluzone® Quadrivalent Group (N=1217)
Upper respiratory tract infection (Infections and infestations) | 111 | 102
Cough (Respiratory, thoracic and mediastinal disorders) | 70 | 77
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 59 | 76
Nasopharyngitis (Infections and infestations) | 66 | 54
Diarrhoea (Gastrointestinal disorders) | 66 | 53
Otitis media (Infections and infestations) | 61 | 49
Drowsiness (General disorders) | 471/1159 | 471/1152
Fever (General disorders) | 183/1159 | 178/1152 — During the 7-day post-vaccination period
Irritability/Fussiness (General disorders) | 630/1159 | 582/1152
Loss of Appetite (General disorders) | 391/1159 | 385/1152
Pain (General disorders) | 509/1156 | 462/1151
Fever (General disorders) | 82/1159 | 93/1152 — During the 2-day post-vaccination period

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.